CLINICAL TRIAL: NCT00797875
Title: The Effects of PNF Stretching on Knee Motion Following TKA
Brief Title: PNF Stretching for TKA on ROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chai Huei-Ming, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200803064R
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Total Knee Arthroplasty
Keywords: proprioceptive neuromuscular facilitation stretching technique, total knee arthroplasty, range of motion
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PNF stretching x 5 repetitions for 3 days
  Interventions: Procedure: PNF stretching
- 2 (Active Comparator): passive stretching
  Interventions: Procedure: passive stretching

INTERVENTIONS:
Procedure: PNF stretching — PNF stretching x 5 repetitions and continue 3 days
  Arms: 1
Procedure: passive stretching — passive stretching x 5 repetitions continue 3 days
  Arms: 2

SUMMARY:
To investigate immediate and short term effects on angle of knee flexion, intensity of pain, strength of the knee extensor, and function of the lower extremity by using PNF stretching technique in patients with total knee arthroplasty.

hypothesis:TKA patients may increase ROM after PNF stretching

DETAILED DESCRIPTION:
Proprioceptive neuromuscular facilitation（PNF） is defined as a treatment method that promotes or hastens the response of the neuromuscular mechanism through stimulation of proprioceptors within the related muscles or joints. PNF stretching technique is a therapeutic technique using the PNF concept to the related muslces either to increase neuro-inhibition mechanism for releasing muscle spasm and elongating muscle length, or to increase neuro-excitation mechanism for enhancing muscle strength. Improvement in range of motion using PNF stretching technique has been reported superior to other techniques in previous literature, but those studies have only been done in healthy adults. Less is known in the effect of PNF stretching on improvement in joint restriction. Range of motion limitation usually disturbed the patients with total knee arthroplasty. PNF stretching techniques has been used frequently for patients with total knee arthroplasty in clinical practice to increase range of motion effectively and reduced knee pain during exercise. However there is no evidence-based research in such a technique for patients with total knee arthroplasty. This research project, therefore, will explore application of PNF stretch in changes of knee flexion, pain, muscle strength, and function of the lower extremity following total knee arthroplasty.

Purposes： To investigate immediate and short term effects on angle of knee flexion, intensity of pain, strength of the knee extensor, and function of the lower extremity by using PNF stretching technique in patients with total knee arthroplasty.

Method： Sixty patients who received total knee arthroplasty in National Taiwan University Hospital will be recruited in this study. They will be allocated randomly into either experimental or control groups. Conventional physical therapy will be given to all participants. Besides, the experimental group will assume PNF stretching technique from the third post-operative day to the day of discharge. This technique will be executed by the same physical therapist, including 5 trials of isometric knee extension for 6 s, followed by active knee flexion to the maximum range immediately, and holding for 10s. The rest interval will be 10 s. For the control group, passive stretch technique with the same treatment time will be given, instead. All participants will be asked to do home exercises after discharged from the hospital. The outcome measures will be given before and after the first session treatment on the same day, on the day of discharge, and one month after the operation. The variables measured will be (1) knee flexion angle measured with a universal goniometer, (2) maximum voluntary isometric strength of the knee extensor measured with a hand-held dynamometer, (3) pain score using pain visual analog scale, (4) function performance of the lower extremity measured with timed up and go test, (5) Knee Injury and Osteoarthritis Outcome Score (KOOS) to record 5 dimensions including the symptoms, stiffness, pain, difficulties in knee functions and/or daily activities, limitations in sports or recreational participation, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* OA knee
* primary unilateral TKA

Exclusion Criteria:

* knee flexion>110 or thigh girth > 55 cm
* poor cognition
* CNS or PNS neuromuscular disease
* received operation in recent 3 months
* joint infection and loosening
* revision total knee arthroplasty
* complication during follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
knee flexion angle | baseline and follow up

SECONDARY OUTCOMES:
VAS pain score | baseline and follow up
knee extensor strength | baseline and follow up
time up and go test time | baseline and follow up
KOOS score | baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Ming Chai, PHD, Principal Investigator — Nation Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan